CLINICAL TRIAL: NCT05978401
Title: A Phase I/II Study Evaluating the Safety, Tolerability, and Efficacy of GLS-012 and GLS-010 in Patients With Advanced Non-Small Cell Lung Cancer (Triumph-02)
Brief Title: Safety, Tolerability, and Efficacy of GLS-012 and GLS-010 in Patients With Advanced Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Gloria Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLS-012-21
Record Dates: First submitted 2023-07-26; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Part1 section is a dose-escalation/expansion study in a single-arm setup； Part2 section sets up a control.
Masking Description: Part1 section is a dose-escalation/expansion study in a single-arm setup； Part2 section sets up a control； All processes do not involve blind settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase I Dose-Escalation Stage：GLS-012+GLS-010 (Experimental): Participants will be treated with escalating doses of GLS-010 + GLS-012 to determine the MTD
  Interventions: Drug: GLS-012+GLS-010
- Phase I Expansion Stage：GLS-012+GLS-010 (Experimental): Participants will be enrolled in the expansion stage to better characterize the safety, tolerability, PK variability, and preliminary efficacy of GLS-012+GLS-010 in Advanced Non-Small Cell Lung Cancer.
  Interventions: Drug: GLS-012+GLS-010
- GLS-012+GLS-010+pemetrexed + carboplatin (Experimental): Participants will be enrolled in the expansion stage to better characterize the safety, PK variability, and preliminary efficacy of GLS-012+GLS-010+pemetrexed+carboplatin in Advanced Non-Small Cell Lung Cancer.
  Interventions: Drug: GLS-012+GLS-010+pemetrexed+carboplatin
- GLS-012+GLS-010+paclitaxel+carboplatin (Experimental): Participants will be enrolled in the expansion stage to better characterize the safety, PK variability, and preliminary efficacy of GLS-012+GLS-010+paclitaxel+carboplatin in Advanced Non-Small Cell Lung Cancer.
  Interventions: Drug: GLS-012+GLS-010+paclitaxel+carboplatin

INTERVENTIONS:
Drug: GLS-012+GLS-010 — Two dose levels will be evaluated for GLS-012+GLS-010 administered. GLS-012+GLS-010 will be given via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression or loss of clinical benefit.
  Other Names: LAG3; PD-1
  Arms: Phase I Dose-Escalation Stage：GLS-012+GLS-010
Drug: GLS-012+GLS-010 — Target dose levels will be evaluated for GLS-012+GLS-010 administered. GLS-012+GLS-010 will be given via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression or loss of clinical benefit.
  Other Names: LAG3; PD-1
  Arms: Phase I Expansion Stage：GLS-012+GLS-010
Drug: GLS-012+GLS-010+pemetrexed+carboplatin — GLS-012+GLS-010 will be given via IV infusion on Day 1 of each 21-day cycle in combination with pemetrexed and carboplatin. Combination treatment will be administered 4~6 cycles.GLS-012+GLS-010/GLS-010 may continue until disease progression or loss of clinical benefit.
  Other Names: LAG3; PD-1; chemotherapy
  Arms: GLS-012+GLS-010+pemetrexed + carboplatin
Drug: GLS-012+GLS-010+paclitaxel+carboplatin — GLS-012+GLS-010 will be given via IV infusion on Day 1 of each 21-day cycle in combination with paclitaxel and carboplatin. Combination treatment will be administered 4~6 cycles.GLS-012+GLS-010/GLS-010 may continue until disease progression or loss of clinical benefit.
  Other Names: LAG3; PD-1; chemotherapy
  Arms: GLS-012+GLS-010+paclitaxel+carboplatin

SUMMARY:
This is a multicenter, open Phase I/II study. The trial consists of two parts, Part1 is a dose-escalation/expansion study, Part2 is a combination of GLS-010 and GLS-010+GLS-012 with standard chemotherapy for advanced non-small-cell lung cancer respectively to assess preliminary efficacy at the combination dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects enroll in the study and sign the Informed Consent Form (ICF);
2. Aged ≥18 years and ≤75 years;
3. histologically or cytologically confirmed advanced non-small cell lung cancer without driver genes (diagnostic criteria refer to AJCC 8th edition of squamous or non-squamous non-small cell lung cancer);
4. Subjects with an Eastern Cooperative Oncology Group (ECOG) score of 0 ~1 for physical status;
5. expected survival ≥ 12 weeks;
6. Subjects with measurable lesions (at least 1 extracranial lesion) according to the Solid Tumor Evaluation Criteria (RECIST v1.1).
7. Subjects provide formalin-fixed, paraffin-embedded tumor tissue blocks or unstained tumor specimen sections (at least 6), either archived or freshly obtained within 5 years prior to the first study treatment (freshly obtained is preferred);
8. Organ function meets the following criteria:

   1. Adequate bone marrow reserve (not acceptable for corrective therapy with hematologic products or cell growth factors administered within 14 days prior to first study dose): absolute neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 90 x 109/L, and hemoglobin ≥ 9 g/dL;
   2. Liver: serum albumin ≥ 3.0 g/dL; total bilirubin ≤ 1.5 times the Upper Limit of Normal (ULN), and ALT and AST ≤ 3 times the ULN (or AST and ALT ≤ 5 × ULN for patients with known liver metastases);
   3. Renal: blood creatinine ≤ 1.25 times ULN;
   4. Heart: left ventricular ejection fraction (LVEF) ≥ 50%.
9. Subjects of childbearing potential must be using highly effective contraception during the study and for at least 6 months after the last dose; female subjects of childbearing potential must have a negative blood pregnancy test within 3 days prior to study enrollment.

Exclusion Criteria:

1. Severe immunotherapy-related toxicity during prior treatment with anti-ICIs;
2. Prior grade ≥ 3 irAE on immunotherapy and who have not recovered to grade ≤ 1 from the last adverse reaction to antineoplastic therapy;
3. With primary or secondary immunodeficiency；
4. Any active, known or suspected autoimmune disease;
5. Known CNS metastases ;
6. Prior severe allergic reactions to large protein preparations/monoclonal antibodies (CTCAE V5.0 classification ≥ grade 4);
7. Previous treatment with anti-LAG-3 antibodies;
8. Other malignant tumors within 5 years prior to screening, except cured cervical carcinoma in situ and cured basal cell carcinoma of the skin;
9. Have uncontrolled cardiac clinical symptoms or disease；
10. Subjects have received a live attenuated vaccine (except inactivated viral seasonal influenza vaccine and novel coronavirus vaccine) within 4 weeks prior to the first dose and who will not receive intranasally administered live attenuated influenza vaccine;
11. Pregnant or nursing females；
12. Poorly compliant or otherwise unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
DLT/MTD | 24 months
  To evaluate GLS-012 in combination with GLS-010 dose-limiting toxicity (DLT)/maximum tolerated dose (MTD) in patients with advanced non-small cell lung cancer
Investigator Assessments of Overall Response Rate(ORR) | 24 months
  RECIST v1.1 will be used to determine ORR by investigator

SECONDARY OUTCOMES:
PFS (progression-free survival) | 24 months
  RECIST v1.1 will be used to determine PFS by investigator
Disease Control Rate(DCR) | 24 months
  RECIST v1.1 will be used to determine DCR by investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Shang Hai Pulmonary Hospital, Shanghai, Shanghai Municipality, China